CLINICAL TRIAL: NCT06023719
Title: Multicentric Clinical Investigation To Assess The Safety And Performance Of Disc Care To Prevent Lumbar Disc Herniation Recurrence
Brief Title: Safety And Performance Of Disc Care To Prevent Lumbar Disc Herniation Recurrence
Acronym: ACE-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NEOS Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NEO-RA1-2023-01
Record Dates: First submitted 2023-08-02; First posted 2023-09-05 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Disc Herniation; Disk Herniated Lumbar
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DISC Care (Experimental): DISC Care implant
  Interventions: Device: DISC Care

INTERVENTIONS:
Device: DISC Care — Medical device to prevent disc herniation recurrence
  Other Names: Hernia Blocking System

SUMMARY:
The goal of this clinical investigation is to learn about DISC Care, an Hernia Blocking System, in patients who have undergone lumbar disc hernia surgery. The main questions it aims to answer are:

* if the implant (DISC Care) prevents disc herniation recurrence
* if DISC Care is a safe device

Participants will be implanted with DISC Care and followed up for two years (7 visits).

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 75 years old.
* Posterolateral disc hernia between levels L4 and S1 with radiological (CT scan or MRI) confirmation of neural compression.
* At least six weeks of failed conservative treatment prior to surgery, including physical therapy, use of anti-inflammatory medications at maximum specified dosage and/or administration of epidural/facet injections.
* Minimum posterior disc height of 5 mm at the index level.
* Radiculopathy with positive straight leg raise test.
* ODI score of at least 30/100.
* Subjects who are able to give voluntary informed consent to participate in the clinical investigation and from whom consent has been obtained.
* Subject is able and willing to comply with the protocol requirements.

Exclusion Criteria:

* Spondylolisthesis and/or instability at the index level that, in the judgement of the surgeon, could affect the device implantation.
* Central, foraminal or extraforaminal disc hernia.
* Subject has vertebral bodies of the index level affected by any traumatic, neoplastic, metabolic, or infectious pathology.
* Subject has scoliosis of greater than 20 degrees (both angular and rotational).
* Grossly distorted anatomy due to congenital abnormalities.
* Deformation that affects the posterior corners of the vertebra at the index level (e.g., osteophytes) that, in the judgment of the surgeon, could affect the device implantation.
* Endplate irregularities that, in the judgment of the surgeon, could affect the device implantation.
* Prior surgery at the index lumbar vertebral level that, in the judgment of the surgeon, could affect the device implantation.
* Radiological confirmation of severe facet joint disease or degeneration.
* Patients diagnosed or at a high risk of osteoporosis (such as postmenopausal women and patients receiving long-term treatment with corticosteroids) who present a bone densitometry DXA (dual energy x-ray absorptiometry) T-score of less than -2.0 at the index level.
* Cauda equina syndrome.
* Fever, leucocytosis and/or systemic or localized active infection.
* Systemic inflammation and/or inflammation at the implantation site.
* Any uncontrolled metabolic bone disease that affects the spine.
* Uncontrolled insulin-dependent diabetes mellitus.
* Peripheral neuropathy.
* Active hepatitis, AIDS or HIV.
* Rheumatoid arthritis or other autoimmune disease that affects the spine joints.
* Active or history of any invasive malignancy; patients with curatively-treated malignancies who have been disease-free for at least 5 years are eligible.
* Uncontrolled active tuberculosis or history of uncontrolled tuberculosis in the past 3 years.
* Immunologically suppressed patients.
* Current anticoagulation therapy, unless anticoagulation therapy can be suspended for surgery.
* Patients who have received medication (e.g., methotrexate, alendronate) that interferes with bone mineral metabolism within 4 weeks of the planned date of the index surgery.
* Suspected or known allergies or intolerance to the device materials: titanium, nitinol, stainless steel, polyetheretherketone and polyethylene terephthalate.
* Any condition that precludes the use of general anaesthesia.
* Any condition that precludes the surgical procedure.
* Any contraindication for MRI or CT scan.
* Class III obesity: Body mass index ≥ 40.
* Current alcohol or recreational drug dependency.
* Pregnant or interested in becoming pregnant in the following 24 months.
* Breastfeeding.
* Life expectancy less than 2 years.
* Subject is currently participating or has participated in the previous 4 weeks in any other interventional clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinically symptomatic recurrent lumbar disc herniation | 24 months

SECONDARY OUTCOMES:
Incidence and type of all adverse events (AE) and serious adverse events (SAE). | 6 weeks, 6 months, 12 months, and 24 months
Incidence of clinically asymptomatic recurrent disc herniation | 6 months, 12 months, and 24 months
Incidence of re-interventions | 6 weeks, 6 months, 12 months, and 24 months
Disc height maintenance [mm] related to baseline | 6 months, 12 months, and 24 months
Change in leg and low back pain, related to baseline | 6 weeks, 6 months, 12 months, and 24 months
  0-10 NRS (numeric rating scale)
Change in Low back related disability, related to baseline | 6 weeks, 6 months, 12 months, and 24 months
  Oswestry Disability Index (ODI)
The change in quality of life, compared to baseline | 6 weeks, 6 months, 12 months, and 24 months
  EQ-5D-5L (5-level EQ-5D version)
The change in patient neurological status, compared to baseline | 6 weeks, 6 months, 12 months, and 24 months
  straight leg raise test, reflexes, motor muscle strength and sensory neurological evaluations, classified as normal or abnormal
The degeneration of the disc, in comparison with the preoperative state | 6 months, 12 months, and 24 months
  Pfirrmann intervertebral disc degeneration scale (I, II, III, IV, V)
the direct and indirect costs of the disease and the intervention. | 6 weeks, 6 months, 12 months, and 24 months
  Custom-made questionnaire

OTHER OUTCOMES:
Description of the impact of the procedure (implantation of the device) on the perioperative parameters | Surgery
  Blood loss (mL)
Description of the impact of the procedure (implantation of the device) on the perioperative parameters | Surgery
  X-ray exposition (seconds of x-ray exposition)
Description of the impact of the procedure (implantation of the device) on the perioperative parameters | Surgery
  Surgery duration (minutes)

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital La Princesa, Madrid, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario la Paz, Madrid, Madrid
  - Hospital QuirónSalud Barcelona, Barcelona
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna